CLINICAL TRIAL: NCT00434837
Title: Effects of Initial Graft Tension on Anterior Cruciate Ligament Reconstruction
Brief Title: Initial Graft Tension and ACL Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Braden Fleming, Professor, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01AR047910 (NIH); R01AR047910 (NIH); R01AR074973 (NIH)
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Results first posted 2024-12-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Knee; Ligament; ACL; Reconstruction; Cartilage; Osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-tension (Experimental): Patients recruited to study the initial graft tension during ACL reconstruction surgery who were randomized to the Low-tension group will receive the low-tension treatment with initial graft tension set so that the anterior-posterior (A-P) displacement of the reconstructed knee is equal to that of the uninjured knee.
  Interventions: Procedure: Initial graft tension during ACL reconstruction surgery
- High-tension (Experimental): Patients recruited to study the initial graft tension during ACL reconstruction surgery who were randomized to the High-tension group will receive the high-tension treatment with the initial graft tension set to reduce A-P displacement by 2 millimeters relative to that of the uninjured knee.
  Interventions: Procedure: Initial graft tension during ACL reconstruction surgery
- Uninjured Control Group (No Intervention): Uninjured age, sex, and race matched control group

INTERVENTIONS:
Procedure: Initial graft tension during ACL reconstruction surgery — The amount of tension that is applied to the graft at the time of fixation is being performed with the knee in two different positions. When the knee is at 30 degrees of flexion, the resulting laxity is approximately 2 mm less than the contralateral leg (the "High Tension" treatment). When the tension is performed with the knee in extension (0 degrees of flexion), the the laxity is equal to that of the contralateral leg (the "Low Tension" treatment). Both methods are commonly used in clinical practice. The effect it may have on articular cartilage remains unknown.
  Arms: High-tension; Low-tension

SUMMARY:
The anterior cruciate ligament (ACL) is one of four strong ligaments connecting the bones of the knee joint. If overstretched, the ACL can tear. Reconstruction of a torn ACL is now a common surgical procedure. The amount of tension applied to the ACL during reconstruction may indirectly affect the possible onset of arthritis over time. The purpose of this study is to determine the effect of initial graft tension set during ACL reconstruction surgery on the progression of knee arthritis over at least a 15-year period.

DETAILED DESCRIPTION:
Damage to the ACL is a common injury that usually requires surgical reconstruction to restore function and prevent progression of post-traumatic osteoarthritis. However, the reconstruction procedure frequently causes degenerative changes to the knee joint over time. The amount of tension applied to the ACL during reconstruction may indirectly affect the possible onset of arthritis over time. High tension would result in less joint motion during the initial healing stages, which may make the onset of arthritis less likely. On the other hand, high tension would result in increased compressive forces between the joint surfaces, which could lead to arthritis. The purpose of this study is to evaluate the effect of initial graft tension set during ACL reconstruction surgery on joint cartilage and the development of knee arthritis over at least a 15-year period.

Participants will include candidates for ACL reconstruction surgery using patellar tendon or hamstring tendon grafts. Participants will be randomly assigned to one of two treatment groups:

* Low tension (Group 1) participants will receive low-tension treatment with initial graft tension set so that the anterior-posterior (A-P) displacement of the reconstructed knee is equal to that of the uninjured knee.
* High-tension (Group 2) participants will receive high-tension treatment with initial graft tension set to reduce A-P displacement by 2 millimeters relative to that of the uninjured knee.

Participants will enroll in this 15-year study 1 to 6 weeks prior to ACL surgery. There will be two preoperative study visits: one will include magnetic resonance imaging (MRI) and the other will include a knee evaluation, dynamic function testing, and questionnaires. Postoperative visits occurred immediately following surgery and at 6, 12, 36, 60, 84, 120, 144 and 180 months following surgery. Strength testing, functional testing, x-rays, questionnaires, and a knee exam will occur at most postoperative visits. MRIs will occur at some postoperative visits. An additional group of participants with no evidence of knee injury will serve as a control. The control group will attend all study visits except for the 12-month visit. All participants may be followed for up to 15 years.

ELIGIBILITY:
Inclusion Criteria for Groups 1 and 2:

* ACL injury of only one knee (minor meniscal tears involving less than 1/3 of the meniscus are allowed)
* Candidate for ACL reconstruction surgery using a bone-patellar tendon-bone graft or a four-stranded hamstring tendon graft (looped semitendinosus and gracilis muscles)
* Tegner activity score of 5 or greater, indicating participant is at least moderately active

Exclusion Criteria for Groups 1 and 2:

* ACL tear that has occurred more than 12 months prior to surgery
* Moderate-sized fissures or lesions in knee articular cartilage
* Meniscal tears requiring partial removal of meniscus (tears larger than 1/3 of the meniscus)

Inclusion Criteria for the Control Group:

* Tegner activity score of 5 or greater, indicating participant is at least moderately active

Exclusion Criteria for All Participants:

* Previous injury to either knee
* Increased laxity of the medial collateral ligament (MCL), lateral collateral ligament (LCL), or posterior cruciate ligament (PCL), as compared to the uninjured knee
* Radiographic evidence of degenerative arthritis
* Pregnancy
* Any disease that might place a participant at high risk for articular cartilage damage (e.g., rheumatoid arthritis, osteoporosis, metabolic diseases)

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Braden C. Fleming, PhD, Principal Investigator — Rhode Island Hospital/Brown Medical School
Locations (2):
- United States (2):
  - Rhode Island Hospital/Brown University, Providence, Rhode Island
  - Miriam Hospital/Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon request. Once the study is completed and published, the data records will be made available through ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data are available upon request at any time. There is no end date. Data will also be posted on ClinicalTrials.gov with no end date.
Access Criteria: Available upon request to the PI. Data on ClinicalTrials.gov are publicly available.

REFERENCES:
- [Background] Fleming BC, Hulstyn MJ, Oksendahl HL, Fadale PD. Ligament Injury, Reconstruction and Osteoarthritis. Curr Opin Orthop. 2005 Oct;16(5):354-362. doi: 10.1097/01.bco.0000176423.07865.d2. PMID 17710194
- [Background] Brady MF, Bradley MP, Fleming BC, Fadale PD, Hulstyn MJ, Banerjee R. Effects of initial graft tension on the tibiofemoral compressive forces and joint position after anterior cruciate ligament reconstruction. Am J Sports Med. 2007 Mar;35(3):395-403. doi: 10.1177/0363546506294363. Epub 2007 Jan 11. PMID 17218659
- [Background] Bowers ME, Tung GA, Trinh N, Leventhal E, Crisco JJ, Kimia B, Fleming BC. Effects of ACL interference screws on articular cartilage volume and thickness measurements with 1.5 T and 3 T MRI. Osteoarthritis Cartilage. 2008 May;16(5):572-8. doi: 10.1016/j.joca.2007.09.010. Epub 2007 Oct 22. PMID 17933559
- [Background] Elsaid KA, Fleming BC, Oksendahl HL, Machan JT, Fadale PD, Hulstyn MJ, Shalvoy R, Jay GD. Decreased lubricin concentrations and markers of joint inflammation in the synovial fluid of patients with anterior cruciate ligament injury. Arthritis Rheum. 2008 Jun;58(6):1707-15. doi: 10.1002/art.23495. PMID 18512776
- [Background] Fleming BC, Brady MF, Bradley MP, Banerjee R, Hulstyn MJ, Fadale PD. Tibiofemoral compression force differences using laxity- and force-based initial graft tensioning techniques in the anterior cruciate ligament-reconstructed cadaveric knee. Arthroscopy. 2008 Sep;24(9):1052-60. doi: 10.1016/j.arthro.2008.05.013. Epub 2008 Jun 30. PMID 18760214
- [Background] Bowers ME, Trinh N, Tung GA, Crisco JJ, Kimia BB, Fleming BC. Quantitative MR imaging using "LiveWire" to measure tibiofemoral articular cartilage thickness. Osteoarthritis Cartilage. 2008 Oct;16(10):1167-73. doi: 10.1016/j.joca.2008.03.005. Epub 2008 Apr 14. PMID 18407529
- [Background] Oksendahl HL, Gomez N, Thomas CS, Badger GD, Hulstyn MJ, Fadale PD, Fleming BC. Digital radiographic assessment of tibiofemoral joint space width: a variance component analysis. J Knee Surg. 2009 Jul;22(3):205-12. doi: 10.1055/s-0030-1247750. PMID 19634723
- [Background] Fleming BC, Oksendahl HL, Mehan WA, Portnoy R, Fadale PD, Hulstyn MJ, Bowers ME, Machan JT, Tung GA. Delayed Gadolinium-Enhanced MR Imaging of Cartilage (dGEMRIC) following ACL injury. Osteoarthritis Cartilage. 2010 May;18(5):662-7. doi: 10.1016/j.joca.2010.01.009. Epub 2010 Feb 11. PMID 20188685
- [Background] Mulcahey MK, Monchik KO, Yongpravat C, Badger GJ, Fadale PD, Hulstyn MJ, Fleming BC. Effects of single-bundle and double-bundle ACL reconstruction on tibiofemoral compressive stresses and joint kinematics during simulated squatting. Knee. 2012 Aug;19(4):469-76. doi: 10.1016/j.knee.2011.05.004. Epub 2011 Jun 22. PMID 21696962
- [Background] Miranda DL, Rainbow MJ, Crisco JJ, Fleming BC. Kinematic differences between optical motion capture and biplanar videoradiography during a jump-cut maneuver. J Biomech. 2013 Feb 1;46(3):567-73. doi: 10.1016/j.jbiomech.2012.09.023. Epub 2012 Oct 22. PMID 23084785
- [Background] Miranda DL, Schwartz JB, Loomis AC, Brainerd EL, Fleming BC, Crisco JJ. Static and dynamic error of a biplanar videoradiography system using marker-based and markerless tracking techniques. J Biomech Eng. 2011 Dec;133(12):121002. doi: 10.1115/1.4005471. PMID 22206419
- [Background] Bowers ME, Tung GA, Oksendahl HL, Hulstyn MJ, Fadale PD, Machan JT, Fleming BC. Quantitative magnetic resonance imaging detects changes in meniscal volume in vivo after partial meniscectomy. Am J Sports Med. 2010 Aug;38(8):1631-7. doi: 10.1177/0363546510364054. Epub 2010 May 4. PMID 20442327
- [Background] Coats-Thomas MS, Miranda DL, Badger GJ, Fleming BC. Effects of ACL reconstruction surgery on muscle activity of the lower limb during a jump-cut maneuver in males and females. J Orthop Res. 2013 Dec;31(12):1890-6. doi: 10.1002/jor.22470. Epub 2013 Aug 21. PMID 23966333
- [Background] Rainbow MJ, Miranda DL, Cheung RT, Schwartz JB, Crisco JJ, Davis IS, Fleming BC. Automatic determination of an anatomical coordinate system for a three-dimensional model of the human patella. J Biomech. 2013 Aug 9;46(12):2093-6. doi: 10.1016/j.jbiomech.2013.05.024. Epub 2013 Jun 20. PMID 23791087
- [Background] Miranda DL, Fadale PD, Hulstyn MJ, Shalvoy RM, Machan JT, Fleming BC. Knee biomechanics during a jump-cut maneuver: effects of sex and ACL surgery. Med Sci Sports Exerc. 2013 May;45(5):942-51. doi: 10.1249/MSS.0b013e31827bf0e4. PMID 23190595
- [Background] Zandiyeh P, Parola LR, Fleming BC, Beveridge JE. Wavelet analysis reveals differential lower limb muscle activity patterns long after anterior cruciate ligament reconstruction. J Biomech. 2022 Mar;133:110957. doi: 10.1016/j.jbiomech.2022.110957. Epub 2022 Jan 20. PMID 35114581
- [Background] Behnke AL, Parola LR, Karamchedu NP, Badger GJ, Fleming BC, Beveridge JE. Neuromuscular function in anterior cruciate ligament reconstructed patients at long-term follow-up. Clin Biomech (Bristol). 2021 Jan;81:105231. doi: 10.1016/j.clinbiomech.2020.105231. Epub 2020 Nov 17. PMID 33246796
- [Background] Zandiyeh P, Parola LR, Costa MQ, Hague MJ, Molino J, Fleming BC, Beveridge JE. Long-Term Bilateral Neuromuscular Function and Knee Osteoarthritis after Anterior Cruciate Ligament Reconstruction. Bioengineering (Basel). 2023 Jul 6;10(7):812. doi: 10.3390/bioengineering10070812. PMID 37508839
- [Result] Fleming BC, Fadale PD, Hulstyn MJ, Shalvoy RM, Oksendahl HL, Badger GJ, Tung GA. The effect of initial graft tension after anterior cruciate ligament reconstruction: a randomized clinical trial with 36-month follow-up. Am J Sports Med. 2013 Jan;41(1):25-34. doi: 10.1177/0363546512464200. Epub 2012 Nov 9. PMID 23144370
- [Result] Akelman MR, Fadale PD, Hulstyn MJ, Shalvoy RM, Garcia A, Chin KE, Duryea J, Badger GJ, Tung GA, Fleming BC. Effect of Matching or Overconstraining Knee Laxity During Anterior Cruciate Ligament Reconstruction on Knee Osteoarthritis and Clinical Outcomes: A Randomized Controlled Trial With 84-Month Follow-up. Am J Sports Med. 2016 Jul;44(7):1660-70. doi: 10.1177/0363546516638387. Epub 2016 Apr 19. PMID 27159308
- [Result] Biercevicz AM, Akelman MR, Fadale PD, Hulstyn MJ, Shalvoy RM, Badger GJ, Tung GA, Oksendahl HL, Fleming BC. MRI volume and signal intensity of ACL graft predict clinical, functional, and patient-oriented outcome measures after ACL reconstruction. Am J Sports Med. 2015 Mar;43(3):693-9. doi: 10.1177/0363546514561435. Epub 2014 Dec 24. PMID 25540298
- [Result] Ware JK, Owens BD, Akelman MR, Karamchedu NP, Fadale PD, Hulstyn MJ, Shalvoy RM, Badger GJ, Fleming BC. Preoperative KOOS and SF-36 Scores Are Associated With the Development of Symptomatic Knee Osteoarthritis at 7 Years After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2018 Mar;46(4):869-875. doi: 10.1177/0363546517751661. Epub 2018 Feb 5. PMID 29401408
- [Result] DeFroda SF, Karamchedu NP, Owens BD, Bokshan SL, Sullivan K, Fadale PD, Hulstyn MJ, Shalvoy RM, Badger GJ, Fleming BC. Tibial tunnel widening following anterior cruciate ligament reconstruction: A retrospective seven-year study evaluating the effects of initial graft tensioning and graft selection. Knee. 2018 Dec;25(6):1107-1114. doi: 10.1016/j.knee.2018.08.003. Epub 2018 Nov 7. PMID 30414786
- [Result] Kiapour AM, Yang DS, Badger GJ, Karamchedu NP, Murray MM, Fadale PD, Hulstyn MJ, Shalvoy RM, Fleming BC. Anatomic Features of the Tibial Plateau Predict Outcomes of ACL Reconstruction Within 7 Years After Surgery. Am J Sports Med. 2019 Feb;47(2):303-311. doi: 10.1177/0363546518823556. Epub 2019 Jan 14. PMID 30640519
- [Result] Fleming BC, Fadale PD, Hulstyn MJ, Shalvoy RM, Tung GA, Badger GJ. Long-term outcomes of anterior cruciate ligament reconstruction surgery: 2020 OREF clinical research award paper. J Orthop Res. 2021 May;39(5):1041-1051. doi: 10.1002/jor.24794. Epub 2020 Jul 17. PMID 32639610
- [Result] DeFroda SF, Karamchedu NP, Budacki R, Wiley T, Fadale PD, Hulstyn MJ, Shalvoy RM, Badger GJ, Fleming BC, Owens BD. Evaluation of Graft Tensioning Effects in Anterior Cruciate Ligament Reconstruction between Hamstring and Bone-Patellar Tendon Bone Autografts. J Knee Surg. 2021 Jun;34(7):777-783. doi: 10.1055/s-0039-3402046. Epub 2020 Jan 21. PMID 31962350
- [Result] Costa MQ, Badger GJ, Chrostek CA, Carvalho OD, Faiola SL, Fadale PD, Hulstyn MJ, Gil HC, Shalvoy RM, Fleming BC. Effects of Initial Graft Tension and Patient Sex on Knee Osteoarthritis Outcomes After ACL Reconstruction: A Randomized Controlled Clinical Trial With 10- to 12-Year Follow-up. Am J Sports Med. 2022 Nov;50(13):3510-3521. doi: 10.1177/03635465221124917. Epub 2022 Oct 19. PMID 36259724
- [Result] Breker AN, Badger GJ, Kiapour AM, Costa MQ, Fleming EN, Ferrara SL, Chrostek CA, Fadale PD, Hulstyn MJ, Shalvoy RM, Gil HC, Fleming BC. Effect of Initial Graft Tension on Knee Osteoarthritis Outcomes After ACL Reconstruction: A Randomized Controlled Clinical Trial With 15-Year Follow-up. Orthop J Sports Med. 2025 Mar 4;13(3):23259671251320972. doi: 10.1177/23259671251320972. eCollection 2025 Mar. PMID 40052176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between February 2004 and February 2007 in clinics of participating doctors: Dr. Paul D. Fadale, Dr. Michael J. Hulstyn, and Dr. Robert M. Shalvoy.
Pre-assignment Details: Patients between the age of 15-50 with isolated unilateral ACL injuries were considered for eligibility. Patients were excluded from the study if they required meniscectomy greater than 1/3 of meniscus, showed increased laxity of knee ligaments, or had a history of previous knee injuries and/or developing osteoarthritis.
  Of 108 subjects initially recruited to tension groups, 18 were excluded pre- or during surgery.
Period: Overall Study
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Started | 46 | 44 | 60
6 Months | 39 | 37 | 0
1 Year | 35 | 34 | 48
3 Years | 44 | 41 | 48
7 Years | 36 | 36 | 34
10-12 Years | 32 | 28 | 35
Completed | 26 | 21 | 30
Not Completed | 20 | 23 | 30
Not completed — Lost to Follow-up | 20 | 23 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-tension | High-tension | Uninjured Control Group | Total
Number analyzed (Participants) | 46 | 44 | 60 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (9.26) | 23.1 (7.19) | 25.3 (6.15) | 24.2 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 26 | 74
  Male | 24 | 18 | 34 | 76
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43 | 36 | 52 | 131
  Black | 0 | 2 | 1 | 3
  Asian | 0 | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  More than one race | 0 | 1 | 0 | 1
  Hispanic or Latino | 2 | 3 | 3 | 8
  Unknown/Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 46 | 44 | 60 | 150
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.7 (3.20) | 24.5 (3.56) | 23.9 (3.14) | 24.3 (3.28)
Time from injury to surgery [Mean (Standard Deviation); unit: days] — Population: Control subjects did not undergo ACL reconstruction and were not included in the calculations.
  5 patients in the high-tension group and 1 patient in the low-tension group did not report an exact injury date and are excluded from this variable.
  days
    number analyzed (Participants) | 45 | 39 | 0 | 84
    (all) | 112 (86.5) | 116 (119) |  | 114 (102)
Graft type [Count of Participants; unit: Participants] — Population: Control patients did not undergo ACL reconstruction and therefore were not assigned a graft type.
  Participants
    number analyzed (Participants) | 46 | 44 | 0 | 90
    Autologous Patellar Tendon | 31 | 27 |  | 58
    Autologous Hamstring Tendon | 15 | 17 |  | 32

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Joint Space Narrowing (Midpoint Method)
Description: Medial joint space width measurements were obtained from radiographs preoperatively and postoperatively using the semiflexed metatarsophalangeal view. Radiographs were taken of each knee, and the medial compartment joint space width was measured by calculating the distance between the femoral and tibial intersections with the bisecting midpoint line. Analysis was conducted using a MATLAB program. (Mehta N, Duryea J, Badger GJ, et al. Comparison of 2 Radiographic Techniques for Measurement of Tibiofemoral Joint Space Width. Orthop J Sports Med. 2017;5(9):2325967117728675. Published 2017 Sep 26. doi:10.1177/2325967117728675) Subjects are identified as having radiographic signs of OA if they exhibit a change in the medial or lateral compartments greater than 0.30 mm over the study period.
  This was the first method used for the study. It was used for baseline and 3-year follow-up prior to switching to the 'surface-fit' method at the 7-year follow-up.
Time Frame: 3 years
Population: Insufficient time for imaging; loss to follow-up.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
mm
  Baseline: number analyzed (Participants) | 45 | 44 | 58
  Baseline | 0.0613 [-0.1640 to 0.2870] | 0.0634 [-0.1260 to 0.2530] | -0.0321 [-0.1850 to 0.1210]
  1-year: number analyzed (Participants) | 38 | 37 | 46
  1-year | 0.1374 [-0.0420 to 0.3170] | 0.1941 [0.0342 to 0.3540] | -0.2413 [-0.4090 to -0.0740]
  3-years: number analyzed (Participants) | 34 | 34 | 36
  3-years | 0.0705 [-0.0700 to 0.2110] | 0.0192 [-0.1200 to 0.1580] | -0.1321 [-0.3220 to 0.0575]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 3-year analysis; Test type: Superiority; p = .27, ANOVA

2. Primary Outcome: Radiographic Joint Space Narrowing (Surface-Fit Method)
Description: Medial joint space width measurements were obtained from radiographs preoperatively and postoperatively using the semiflexed metatarsophalangeal view. Radiographs were taken of each knee, and the medial compartment joint space width was measured at the midline of the compartment in the coronal plane using a validated computer algorithm.
  (Duryea et al., Trainable rule-based algorithm for the measurement of joint space width in digital radiographic images of the knee, Medical Physics 27, 580 (2000); doi: 10.1118/1.598897). Subjects are identified as having radiographic signs of OA if they exhibit a change in the medial or lateral compartments greater than 0.30mm over the study period.
  The surface-fit method was used for the 7-year follow-up and baseline radiographs instead of the Midpoint Method, after confirming less variability across knees within a participant. (Mehta et al. 2017)
Time Frame: 7 years
Population: Insufficient time for imaging; loss to follow-up. Baseline images of subjects presented at 7-year follow-up were analyzed again retroactively with this method.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
mm
  Baseline: number analyzed (Participants) | 23 | 21 | 24
  Baseline | 0.1483 [-0.0979 to 0.3944] | 0.0029 [-0.2001 to 0.2058] | -0.0492 [-0.2041 to 0.1058]
  7-years: number analyzed (Participants) | 19 | 16 | 21
  7-years | 0.1858 [-0.0370 to 0.4086] | 0.1969 [-0.0855 to 0.4792] | -0.2314 [-0.4259 to -0.0369]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 7-year analysis; Test type: Superiority; p = .08, ANOVA

3. Primary Outcome: Radiographic Joint Space Narrowing (Kiapour Method)
Description: Joint space width measurements in the medial compartment were calculated from weightbearing radiographs using the semi-flexed metatarsophalangeal view. Radiographs were manually segmented to outline articular surfaces of femur and tibia using Mimics. A custom program in MATLAB developed by Dr. Ata Kiapour was used to calculate joint space width as the perpendicular distance between the femoral condyle and tibial plateau boundaries at 25% of total bicondylar width. Measured JSW values were then scaled using image distances between beads of a calibration standard taped to the fibular head.
  This method was used for the baseline, 10-12, and 15-year follow-up as a comparable in-house method to the surface-fit method.
  Subjects are identified as having radiographic signs of OA if they exhibit a change in the medial or lateral compartments greater than 0.30 mm over the study period.
Time Frame: 15 years
Population: Insufficient time for imaging; loss to follow-up. Method was used retroactively for existing baseline images.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
mm
  Baseline: number analyzed (Participants) | 45 | 44 | 60
  Baseline | -0.1076 [-0.3421 to 0.1268] | 0.0653 [-0.1947 to 0.3254] | -0.0876 [-0.3242 to 0.1490]
  10-12-year: number analyzed (Participants) | 26 | 21 | 26
  10-12-year | -0.1038 [-0.6593 to 0.4516] | 0.3238 [-0.0686 to 0.7162] | 0.3269 [-0.1281 to 0.7819]
  15-year: number analyzed (Participants) | 16 | 12 | 18
  15-year | 0.1136 [-0.5391 to 0.7664] | 0.5509 [-0.1457 to 1.2474] | -0.1553 [-0.5961 to 0.2856]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .22, ANOVA

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Symptoms
Description: The five dimensions of Knee Osteoarthritis Outcome Score were scored separately: pain , symptoms ,activities of daily life function, sport and recreation function, and knee-related quality of life . Each sub score has a 0-100 scale. 0- extreme knee problems and 100- no knee problems.
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the symptoms score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 70.3704 [65.6310 to 75.1100] | 70.4319 [65.0120 to 75.8520] | 96.7292 [95.6970 to 97.7560]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 79.5168 [75.6389 to 83.3947] | 78.4184 [72.0655 to 84.7712] |
  1-year: number analyzed (Participants) | 36 | 39 | 47
  1-year | 84.1270 [80.1998 to 88.0542] | 80.0824 [75.0444 to 85.1205] | 95.8207 [94.4758 to 97.1655]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 85.9073 [81.9161 to 89.8986] | 82.1429 [76.7482 to 87.5375] | 93.2234 [90.4490 to 95.9979]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 82.2421 [76.9068 to 87.5773] | 85.8135 [80.5316 to 91.0954] | 92.3319 [89.4216 to 95.2423]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 83.4110 [77.9542 to 88.8677] | 85.0257 [78.8811 to 91.1703] | 91.7351 [89.1559 to 94.3144]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 84.2033 [78.8341 to 89.5725] | 83.1633 [77.3211 to 89.0054] | 92.6190 [89.0315 to 96.2066]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .0078, ANOVA

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Pain
Description: as for outcome 4
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the pain score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 75.3549 [70.8954 to 79.8145] | 77.0187 [72.5225 to 81.5150] | 98.8889 [98.3103 to 99.4675]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 86.6422 [83.0298 to 90.2545] | 86.2302 [80.3802 to 92.0801] |
  1-year: number analyzed (Participants) | 36 | 39 | 47
  1-year | 90.2317 [86.8120 to 93.6510] | 88.9245 [85.2901 to 92.5589] | 98.1679 [97.1089 to 99.2268]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 90.6907 [86.8264 to 94.5549] | 91.0948 [87.6175 to 94.5720] | 96.2963 [93.7527 to 98.8400]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 90.5671 [86.6955 to 94.4387] | 92.8241 [89.0008 to 96.6474] | 96.3848 [94.5122 to 98.2574]
  10-12-years: number analyzed (Participants) | 31 | 27 | 35
  10-12-years | 90.8606 [87.1920 to 94.5293] | 91.0493 [85.7998 to 96.2987] | 97.3806 [95.8193 to 98.9419]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 90.7051 [86.6543 to 94.7559] | 93.5185 [89.9347 to 97.1023] | 98.1481 [96.6234 to 99.6729]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .0018, ANOVA

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Activities of Daily Life
Description: as for outcome 4
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the ADL score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 85.7680 [81.4825 to 90.0534] | 84.3365 [80.3405 to 88.3326] | 99.9755 [99.9265 to 100.0245]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 94.8097 [92.8513 to 96.7681] | 90.5462 [84.5811 to 96.5114] |
  1-year: number analyzed (Participants) | 36 | 39 | 47
  1-year | 94.5440 [91.6380 to 97.45] | 95.0415 [92.5158 to 97.5672] | 99.5037 [99.1101 to 99.9513]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 94.5151 [91.4240 to 97.6062] | 95.8478 [93.4576 to 98.2379] | 98.6779 [97.3206 to 100.0352]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 94.8938 [91.7594 to 98.0282] | 96.5686 [93.5857 to 99.5515] | 98.6592 [97.7352 to 99.5832]
  10-12-years: number analyzed (Participants) | 31 | 27 | 35
  10-12-years | 95.7313 [93.0805 to 98.3821] | 94.2263 [89.7832 to 98.6694] | 99.4094 [98.9962 to 99.8226]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 94.4005 [90.7854 to 98.0155] | 97.6190 [95.4553 to 99.7827] | 99.0686 [98.2595 to 99.8778]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .015, ANOVA

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Sport
Description: as for outcome 4
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the sport score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 41 | 41 | 59
  Baseline | 54.7866 [47.7469 to 61.8263] | 54.8882 [47.9207 to 61.8557] | 98.0720 [96.9090 to 99.2351]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 75.7059 [69.6028 to 81.8090] | 73.9286 [67.9167 to 79.9404] |
  1-year: number analyzed (Participants) | 36 | 39 | 47
  1-year | 79.5708 [74.4160 to 84.7260] | 80.3846 [74.3300 to 86.4392] | 95.9575 [93.5311 to 98.3838]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 81.6216 [76.0324 to 87.2108] | 83.2353 [77.2962 to 89.1744] | 92.6923 [87.0987 to 98.2859]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 80.0000 [73.6754 to 86.3246] | 87.7778 [82.1937 to 93.3618] | 93.6765 [90.1870 to 97.1659]
  10-12-years: number analyzed (Participants) | 31 | 27 | 35
  10-12-years | 85.0000 [79.8987 to 90.1013] | 85.7407 [78.9669 to 92.5146] | 94.0000 [90.7910 to 97.2090]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 80.5769 [71.9835 to 89.1703] | 87.3810 [81.9653 to 92.7966] | 95.0000 [91.2021 to 98.7979]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .003, ANOVA

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) - Quality of Life
Description: as for outcome 4
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the QOL score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 59
  Baseline | 35.6944 [30.6595 to 40.7294] | 37.9360 [31.5675 to 44.3046] | 97.3517 [95.4119 to 99.2915]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 61.2132 [54.8600 to 67.5665] | 58.1250 [52.2390 to 64.0110] |
  1-year: number analyzed (Participants) | 36 | 39 | 47
  1-year | 74.0612 [68.7190 to 79.4040] | 67.6282 [60.4756 to 74.7808] | 95.4122 [92.1426 to 98.6819]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 78.8851 [71.6463 to 86.1239] | 77.7674 [71.2467 to 84.2680] | 93.2692 [88.3153 to 98.2231]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 75.6944 [68.8883 to 82.5006] | 81.2500 [73.6973 to 88.8027] | 92.4632 [87.5754 to 97.3511]
  10-12-years: number analyzed (Participants) | 31 | 27 | 35
  10-12-years | 85.2823 [79.8469 to 90.7176] | 77.7778 [68.4543 to 87.1013] | 94.2857 [90.7215 to 97.8499]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 81.9712 [75.1476 to 88.7947] | 75.5952 [64.3980 to 86.7924] | 94.7917 [91.0095 to 98.5739]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .0006, ANOVA

9. Secondary Outcome: Knee Joint Laxity
Description: Difference in Anterior-Posterior (A-P) knee laxity value; A-P laxity is defined as the amount of A-P directed translation of the tibia (relative to the femur) between the shear load limits of -90 N (posterior) and 133 N (anterior).
Time Frame: 15 years
Population: Loss to follow-up or questionnaire-only participant
Measure: Mean (95% Confidence Interval); unit: Millimeters
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
Millimeters
  Baseline | 4.5107 [3.8889 to 5.1324] | 4.1532 [3.3972 to 4.9091] | 0.4383 [0.1187 to 0.7580]
  6-months: number analyzed (Participants) | 38 | 36 | 0
  6-months | 1.6605 [0.8297 to 2.4914] | 0.8389 [-0.1027 to 1.7805] |
  1-year: number analyzed (Participants) | 39 | 37 | 48
  1-year | 2.3026 [1.4965 to 3.1086] | 2.1378 [1.1908 to 3.0848] | 0.1417 [-0.2299 to 0.5133]
  3-years: number analyzed (Participants) | 33 | 33 | 37
  3-years | 1.7727 [1.0241 to 2.5213] | 2.4545 [1.5927 to 3.3164] | -0.8919 [-1.4717 to -0.3121]
  7-years: number analyzed (Participants) | 31 | 29 | 32
  7-years | 1.3436 [-0.2096 to 2.8969] | 1.3890 [0.2023 to 2.5756] | -0.3301 [-1.2242 to 0.5641]
  10-12-years: number analyzed (Participants) | 26 | 21 | 28
  10-12-years | 1.0763 [-0.3137 to 2.4662] | 1.7086 [-0.2736 to 3.6909] | -0.0328 [-0.9127 to 0.8470]
  15-years: number analyzed (Participants) | 18 | 12 | 19
  15-years | .9907 [0.3171 to 1.6644] | 1.5967 [-0.8270 to 4.0204] | 1.1002 [-0.4689 to 1.5917]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .15, ANOVA

10. Secondary Outcome: Limb Strength International Knee Documentation Committee (IKDC) Score
Description: Clinical outcome was assessed using the 2000 IKDC Knee Examination Score (http://www.sportsmed.org). The IKDC scores evaluate 4 categories: function, symptoms, range of knee motion, and clinical examination.The IKDC score rates knees as normal (A), nearly normal (B), abnormal (C), and severely abnormal (D), with the final IKDC rating based on the score of the worst category.
Time Frame: 15 years
Population: Loss to follow-up or questionnaire-only subject
Measure: Count of Participants; unit: Participants
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
Participants
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline: A | 0 | 0 | 58
  Baseline: B | 27 | 28 | 2
  Baseline: C | 17 | 13 | 0
  Baseline: D | 1 | 2 | 0
  6-months: number analyzed (Participants) | 39 | 37 | 0
  6-months: A | 21 | 21 |
  6-months: B | 16 | 15 |
  6-months: C | 2 | 1 |
  6-months: D | 0 | 0 |
  1-year: number analyzed (Participants) | 37 | 37 | 48
  1-year: A | 21 | 16 | 46
  1-year: B | 11 | 16 | 2
  1-year: C | 5 | 5 | 0
  1-year: D | 0 | 0 | 0
  3-years: number analyzed (Participants) | 33 | 33 | 37
  3-years: A | 17 | 17 | 30
  3-years: B | 12 | 11 | 5
  3-years: C | 4 | 5 | 2
  3-years: D | 0 | 0 | 0
  7-years: number analyzed (Participants) | 32 | 29 | 32
  7-years: A | 9 | 7 | 24
  7-years: B | 16 | 22 | 8
  7-years: C | 7 | 0 | 0
  7-years: D | 0 | 0 | 0
  10-12-years: number analyzed (Participants) | 26 | 22 | 27
  10-12-years: A | 6 | 8 | 22
  10-12-years: B | 19 | 9 | 4
  10-12-years: C | 1 | 3 | 0
  10-12-years: D | 0 | 2 | 1
  15-years: number analyzed (Participants) | 18 | 13 | 20
  15-years: A | 8 | 5 | 14
  15-years: B | 6 | 6 | 5
  15-years: C | 3 | 2 | 0
  15-years: D | 1 | 0 | 1
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .34, Chi-squared

11. Secondary Outcome: Short Form-36 (SF-36) Health Survey Physical Functioning
Description: The SF-36 evaluates general health related to physical function, role limitations, bodily pain, vitality, social functioning, mental health, and health transition. Each sub score is on a 0-100 scale. 100 indicates no problems and 0 indicates severe problems.
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the physical functioning score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 70.0000 [64.2149 to 75.7851] | 70.1163 [64.3606 to 75.8719] | 98.3333 [96.3071 to 100.3595]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 83.8971 [78.7746 to 89.0195] | 83.1429 [78.7302 to 87.5555] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 89.1667 [85.3313 to 93.0021] | 90.7500 [87.7613 to 93.7387] | 99.0426 [98.0704 to 100.0148]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 89.9865 [84.6607 to 95.3123] | 93.9706 [91.2091 to 96.7320] | 95.8974 [91.7759 to 100.0189]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 91.9444 [88.5808 to 95.2081] | 95.1389 [91.9395 to 98.3382] | 97.6471 [94.6546 to 100.6395]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 90.0000 [83.9539 to 96.0461] | 95.1786 [91.7421 to 98.6151] | 96.4286 [92.4601 to 100.3970]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 91.1538 [86.9444 to 95.3633] | 91.9048 [82.6185 to 101.1911] | 97.1667 [94.9914 to 99.3420]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .17, ANOVA

12. Secondary Outcome: Short Form-36 (SF-36) Health Survey Physical Role
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the physical role score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 59.5833 [51.3374 to 67.8293] | 54.0698 [45.2521 to 62.8874] | 97.6389 [95.1465 to 100.1313]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 86.3971 [79.9905 to 92.8036] | 82.5840 [75.5790 to 89.5890] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 91.8403 [86.1108 to 97.5697] | 92.0313 [85.7822 to 98.2803] | 96.4096 [92.5422 to 100.2769]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 91.7230 [84.9064 to 98.5395] | 96.6912 [93.2614 to 100.1210] | 95.6731 [91.6396 to 99.7066]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 94.2708 [90.5649 to 97.9767] | 97.5694 [94.5699 to 100.5690] | 96.5074 [92.1493 to 100.8654]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 96.5276 [94.1733 to 98.9719] | 96.2054 [92.0099 to 100.4008] | 95.7143 [91.4009 to 100.0276]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 90.1442 [83.1057 to 97.1827] | 96.1310 [90.3370 to 101.9249] | 95.2083 [91.4460 to 98.9706]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .25, ANOVA

13. Secondary Outcome: Short Form-36 (SF-36) Health Survey General Health
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the general health score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 81.9111 [77.6502 to 86.1720] | 84.9767 [80.9132 to 89.0403] | 86.1667 [83.4506 to 88.8828]
  6 months: number analyzed (Participants) | 36 | 36 | 0
  6 months | 83.4412 [79.0232 to 87.8592] | 82.2286 [76.7705 to 87.6867] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 84.9722 [81.3926 to 88.5519] | 85.6750 [81.9283 to 89.4217] | 86.6170 [82.9112 to 90.3228]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 82.4865 [77.9758 to 86.9972] | 85.2941 [80.2182 to 90.3700] | 85.1795 [81.2033 to 89.1557]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 80.1111 [75.1838 to 85.0384] | 84.8611 [79.9965 to 89.7257] | 86.6765 [82.9893 to 90.3636]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 81.9355 [76.5530 to 87.3180] | 82.3214 [75.8139 to 88.8290] | 84.2000 [80.0826 to 88.3174]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 80.8462 [75.0572 to 86.6351] | 84.7143 [79.5080 to 89.9205] | 82.4655 [77.3330 to 87.5981]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .61, ANOVA

14. Secondary Outcome: Short Form-36 (SF-36) Health Survey Bodily Pain
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the bodily pain score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 62.3778 [56.8292 to 67.9264] | 61.0000 [54.3793 to 67.6207] | 86.6500 [83.3107 to 89.9893]
  6 months: number analyzed (Participants) | 36 | 35 | 0
  6 months | 80.2727 [75.5851 to 84.9603] | 77.5571 [70.8949 to 84.2194] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 82.4167 [76.0573 to 88.7760] | 85.1750 [80.1712 to 90.1788] | 87.0000 [82.5563 to 91.4437]
  3-years: number analyzed (Participants) | 37 | 34 | 38
  3-years | 84.6216 [78.1458 to 91.0974] | 86.8824 [81.8599 to 91.9048] | 84.7895 [79.7484 to 89.8305]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 79.2778 [73.5094 to 85.0461] | 86.8611 [81.4491 to 92.2731] | 86.0000 [81.7511 to 90.2489]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 83.1613 [77.3399 to 88.9827] | 88.1786 [82.4937 to 93.8634] | 82.4857 [75.4688 to 89.5027]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 78.4231 [70.1272 to 86.7190] | 89.1743 [82.8574 to 96.5712] | 81.6667 [73.5097 to 89.8237]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .15, ANOVA

15. Secondary Outcome: Short Form-36 (SF-36) Health Survey Vitality
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the vitality score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 62.6733 [57.8691 to 67.4776] | 64.0988 [58.4637 to 69.7340] | 73.2292 [70.0119 to 76.4464]
  6 months: number analyzed (Participants) | 36 | 35 | 0
  6 months | 65.3409 [59.6212 to 71.0606] | 73.3929 [67.5268 to 79.2589] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 69.7917 [64.4566 to 75.1268] | 71.4063 [65.6558 to 77.1567] | 70.3457 [66.8020 to 73.8895]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 69.2568 [64.2376 to 74.2759] | 73.1618 [68.4258 to 77.8977] | 73.5577 [69.5687 to 77.5467]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 68.4028 [62.0262 to 74.7794] | 72.9456 [67.5190 to 78.3722] | 70.9559 [66.0367 to 75.8751]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 67.4058 [61.6264 to 73.1852] | 72.3214 [64.6712 to 79.9716] | 70.0000 [65.7744 to 74.2256]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 64.9038 [59.0560 to 70.7517] | 70.5357 [61.8531 to 79.2184] | 67.9167 [61.2949 to 74.5384]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .53, ANOVA

16. Secondary Outcome: Short Form-36 (SF-36) Health Survey Social Function
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the social function score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 81.1111 [74.9987 to 87.2235] | 75.5814 [68.6177 to 82.5451] | 96.4583 [94.2723 to 98.6443]
  6 months: number analyzed (Participants) | 36 | 35 | 0
  6 months | 88.6364 [82.6564 to 94.6164] | 90.0000 [83.5211 to 96.4789] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 92.7083 [87.8893 to 97.5274] | 92.6563 [86.7899 to 98.5226] | 97.2826 [94.6823 to 99.8829]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 94.5946 [90.5374 to 98.6518] | 97.4265 [94.2990 to 100.5539] | 96.7949 [93.0398 to 100.5500]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 89.9306 [84.4011 to 95.4600] | 96.5278 [93.1338 to 99.9217] | 97.0588 [94.0625 to 100.0552]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 95.9677 [91.8108 to 100.1247] | 96.4286 [92.0894 to 100.7677] | 93.9286 [88.6739 to 99.1833]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 90.3846 [84.9830 to 95.7862] | 92.8571 [84.8970 to 100.8172] | 90.0000 [82.9160 to 97.0840]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .82, ANOVA

17. Secondary Outcome: Short Form-36 (SF-36) Health Survey Emotional Role
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the emotional role score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 85.3704 [79.2249 to 91.5158] | 85.3175 [77.2360 to 93.3989] | 96.6667 [94.3963 to 98.9370]
  6 months: number analyzed (Participants) | 36 | 35 | 0
  6 months | 89.3930 [83.0552 to 95.7308] | 91.9188 [85.9390 to 97.8980] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 92.1278 [86.4565 to 97.7990] | 92.771 [87.0640 to 98.4780] | 98.2277 [96.7422 to 99.7131]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 94.1441 [90.1689 to 98.1194] | 97.5500 [94.6911 to 100.4089] | 96.3667 [92.6007 to 100.1326]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 95.1289 [91.4789 to 98.7985] | 95.6019 [91.4825 to 99.7212] | 97.0588 [93.4789 to 100.6387]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 97.3123 [94.8714 to 99.7531] | 97.3218 [94.4054 to 100.2382] | 97.8571 [94.9122 to 100.8021]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 91.0256 [85.7316 to 96.3197] | 96.8254 [93.7728 to 99.8780] | 97.5000 [94.6516 to 100.3484]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .03, ANOVA

18. Secondary Outcome: Short Form-36 (SF-36) Health Survey Mental Health
Description: as for outcome 11
Time Frame: 15 years
Population: Some subjects omitted responses from questions pertaining to the mental health score. These subjects were omitted from the overall N for score calculations.
  Loss to follow-up between time-points accounts for the remaining population differences. Control subjects were not assessed at 6 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 45 | 43 | 60
  Baseline | 74.1111 [69.6377 to 78.5845] | 74.8837 [69.9327 to 79.8348] | 84.1667 [81.8706 to 86.4628]
  6 months: number analyzed (Participants) | 36 | 35 | 0
  6 months | 80.0000 [74.3068 to 85.6932] | 83.5714 [78.8249 to 88.3180] |
  1-year: number analyzed (Participants) | 36 | 40 | 47
  1-year | 78.4722 [73.0087 to 83.9358] | 82.6250 [77.8140 to 87.4360] | 82.4468 [79.4384 to 85.4552]
  3-years: number analyzed (Participants) | 37 | 34 | 39
  3-years | 82.2973 [78.4693 to 86.1253] | 86.0294 [82.8201 to 89.2387] | 85.5128 [82.6960 to 88.3296]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 79.8611 [74.9900 to 84.7322] | 85.0000 [80.7649 to 89.2352] | 84.8529 [81.7942 to 87.9116]
  10-12-years: number analyzed (Participants) | 31 | 28 | 35
  10-12-years | 80.9677 [76.4137 to 85.5218] | 81.9643 [76.2764 to 87.6522] | 80.7143 [77.3979 to 84.0307]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 78.4135 [74.4059 to 82.4210] | 81.9048 [74.3399 to 89.4696] | 80.6667 [75.4608 to 85.8725]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .67, ANOVA

19. Secondary Outcome: Muscle Atrophy
Description: Thigh circumference 6 cm above the joint line for injured and contralateral knees. Muscle atrophy difference calculated as index-contralateral circumference.
Time Frame: 15 years
Population: Participant population declined due to loss to follow-up or insufficient time to test at the appointment. Control subjects were not tested at the 6-month follow-up.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
centimeters
  Baseline: number analyzed (Participants) | 45 | 43 | 58
  Baseline | -0.0267 [-0.3337 to 0.2803] | -0.2093 [-0.5567 to 0.1381] | 0.0293 [-0.2200 to 0.2785]
  6-months: number analyzed (Participants) | 37 | 35 | 0
  6-months | 0.9324 [0.5463 to 1.3186] | 0.7071 [0.2636 to 1.1507] |
  1-year: number analyzed (Participants) | 38 | 36 | 49
  1-year | 0.6579 [0.3762 to 0.9396] | 0.7896 [0.4142 to 1.1831] | 0.3520 [0.0667 to 0.6374]
  3-years: number analyzed (Participants) | 34 | 33 | 38
  3-years | -0.3359 [-0.6838 to 0.0119] | -0.3030 [-0.6802 to 0.0741] | 0.2105 [-0.0287 to 0.4497]
  7-years: number analyzed (Participants) | 32 | 30 | 31
  7-years | -0.2625 [-0.6054 to 0.0804] | -0.4783 [-0.8105 to -0.1462] | 0.0323 [-0.3045 to 0.3690]
  10-12-years: number analyzed (Participants) | 25 | 22 | 27
  10-12-years | -0.3600 [-0.7333 to 0.0133] | -0.4318 [-0.7151 to -0.1486] | 0.1000 [-0.3127 to 0.5127]
  15-years: number analyzed (Participants) | 17 | 13 | 19
  15-years | -0.2941 [-0.8946 to 0.3063] | -0.7308 [-1.2700 to -0.1916] | 0 [-0.4370 to 0.4370]

20. Secondary Outcome: Whole Organ Magnetic Resonance Image Score (WORMS)
Description: The OA status of the knee was assessed using the semiquantitative Whole Organ Magnetic Resonance Imaging Score (WORMS).The score uses magnetic resonance imaging (MRI) sequences to grade 14 independent features: cartilage signal and morphological characteristics, subarticular bone marrow abnormality, subarticular cysts, subarticular bone attrition, and marginal osteophytes evaluated in 15 regions. The condition of the menisci, cruciate and collateral ligaments, synovitis, loose bodies, and periarticular cysts was also included for a total possible score of 332 points.
  0-indicates no damage in anatomical landmarks assessed. 332-severe damage to the anatomical landmarks assessed.
Time Frame: 15 years
Population: Insufficient time for imaging; loss to follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 17 | 16 | 24
  Baseline | 3.7941 [2.3168 to 5.2714] | 6.1875 [4.1224 to 8.2526] | 0.9167 [-0.2205 to 2.0539]
  1-year: number analyzed (Participants) | 18 | 14 | 24
  1-year | 3.5278 [1.7097 to 5.3459] | 6.9286 [4.3919 to 9.4653] | -0.9583 [-4.3627 to 2.4460]
  3-year: number analyzed (Participants) | 27 | 24 | 12
  3-year | 3.1852 [1.3557 to 5.0146] | 3.2917 [1.0765 to 5.5068] | -0.3333 [-1.5550 to 0.8883]
  7-year: number analyzed (Participants) | 33 | 28 | 31
  7-year | 8.1667 [1.6805 to 14.6528] | 2.8929 [0.2920 to 5.4937] | -1.3548 [-2.7709 to 0.0612]
  10-12-year: number analyzed (Participants) | 26 | 21 | 25
  10-12-year | 11.6731 [2.1720 to 21.1740] | 7.3095 [-0.3080 to 14.9270] | -3.8400 [-9.2980 to 1.6180]
  15-year: number analyzed (Participants) | 15 | 10 | 18
  15-year | 11.2333 [0.6503 to 21.8164] | 10.0000 [-4.1744 to 24.1744] | -1.2500 [-4.5599 to 2.0599]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .051, ANOVA

21. Secondary Outcome: One-legged Hop Test
Description: Ratio of hop distance on the injured knee to the hop distance on the contralateral uninjured knee.
Time Frame: 15 years
Population: Some surgical subjects declined to perform due to knee instability. Other subjects had insufficient time to test. There was loss to follow-up at later timepoints.
Measure: Mean (95% Confidence Interval); unit: percentage of contralateral knee
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
percentage of contralateral knee
  Baseline: number analyzed (Participants) | 45 | 41 | 60
  Baseline | 76.8510 [70.7897 to 82.9124] | 76.9565 [70.8739 to 83.0390] | 101.0724 [99.3010 to 102.8438]
  1-year: number analyzed (Participants) | 43 | 44 | 48
  1-year | 91.2106 [85.9651 to 96.4560] | 93.0460 [89.9935 to 96.0986] | 100.6628 [98.6970 to 102.6287]
  3-years: number analyzed (Participants) | 32 | 32 | 37
  3-years | 94.3962 [91.4571 to 97.3353] | 95.2889 [91.8188 to 98.7590] | 100.7867 [98.5830 to 102.9904]
  7-years: number analyzed (Participants) | 29 | 28 | 31
  7-years | 93.0311 [88.3546 to 97.7075] | 94.8787 [91.2124 to 98.5451] | 101.3066 [98.3556 to 104.2575]
  10-12-years: number analyzed (Participants) | 25 | 22 | 26
  10-12-years | 94.9735 [88.9808 to 100.9663] | 92.2336 [87.4438 to 97.0235] | 100.0648 [96.0300 to 104.0996]
  15-years: number analyzed (Participants) | 17 | 11 | 19
  15-years | 93.2949 [88.3152 to 98.2745] | 85.1336 [64.2280 to 106.0392] | 101.0900 [90.8219 to 111.3570]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results were from the 15-year analysis; Test type: Superiority; p = .14, ANOVA

22. Secondary Outcome: Modified OsteoArthritis Research Society International (OARSI) Score
Description: OARSI-The overall condition of the knee joints of both surgical and contralateral limbs were graded on radiographs by a radiologist. (0-83). 83-severe damage.0- no damage. The difference of the score between surgical and contralateral limbs is also presented.
Time Frame: 15 years
Population: Insufficient time for imaging; loss to follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline: number analyzed (Participants) | 31 | 26 | 31
  Baseline | -0.0541 [-0.2844 to 0.1762] | -0.1081 [-0.3059 to 0.0897] | -0.2604 [-0.7254 to 0.2046]
  1-year: number analyzed (Participants) | 30 | 25 | 28
  1-year | 0 [-0.2300 to 0.2300] | 0.3400 [0.0066 to 0.6730] | -0.3125 [-0.8090 to 0.1840]
  3-year: number analyzed (Participants) | 28 | 24 | 27
  3-year | 0.7679 [0.1160 to 1.7611] | 0.5000 [-0.0370 to 1.0370] | -0.0185 [-0.3270 to 0.2900]
  7-year: number analyzed (Participants) | 30 | 29 | 30
  7-year | 1.0667 [0.1460 to 1.9870] | 0.6724 [0.1930 to 1.1520] | -0.1667 [-0.4340 to 0.1000]
  10-12-year: number analyzed (Participants) | 27 | 21 | 26
  10-12-year | 2.2222 [0.0376 to 4.4070] | 0.7857 [-0.1720 to 1.7430] | -0.0385 [-0.2870 to 0.2100]
  15-year: number analyzed (Participants) | 16 | 12 | 18
  15-year | 2.2813 [-.1722 to 4.7347] | 0.5833 [-0.2276 to 1.3942] | 0.0278 [-0.1063 to 0.1619]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .067, ANOVA

23. Secondary Outcome: Isokinetic Strength
Description: Strength of quadriceps muscles was quantified by averaging the peak torques of 3 repetitions and normalizing these values with respect to body weight.Percent torque of surgical compared to contralateral is presented. If the quadriceps muscle of the surgical limb had the same peak torque as the contralateral, it would be 100%.
Time Frame: 7 years
Population: At baseline, machine measuring isokinetic strength was unavailable for many surgical subjects. Population discrepancies at later time-points include loss to follow-up and machine unavailability. Isokinetic strength was no longer measured after the 7-year follow-up.
Measure: Mean (95% Confidence Interval); unit: percentage of index/contralateral limbs
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
percentage of index/contralateral limbs
  Baseline: number analyzed (Participants) | 9 | 6 | 60
  Baseline | 80.0994 [71.4176 to 88.7811] | 74.6156 [61.9163 to 87.3148] | 101.8830 [98.8688 to 104.8972]
  1-year: number analyzed (Participants) | 35 | 34 | 48
  1-year | 86.6887 [81.0567 to 92.3206] | 82.6245 [76.9096 to 88.3393] | 105.7979 [102.8176 to 108.7783]
  3-years: number analyzed (Participants) | 32 | 31 | 38
  3-years | 94.4971 [89.0526 to 98.0987] | 94.4971 [89.4719 to 99.5223] | 102.3595 [94.9144 to 109.8046]
  7-years: number analyzed (Participants) | 28 | 26 | 29
  7-years | 99.6495 [90.9347 to 108.3642] | 103.1218 [95.6583 to 110.5853] | 99.9448 [95.3044 to 104.5852]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results were from the 7-year analysis; Test type: Superiority; p = .54, ANOVA

24. Secondary Outcome: Tegner Activity Scale
Description: The Tegner activity scale graded activity level based on work and sports activity on a scale of 1-10 with 1 representing physical disability due to knee problems and 10 indicating national or international level soccer participation.
Time Frame: 15-years
Population: Subjects were lost to follow-up throughout the study.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Low-tension | High-tension | Uninjured Control Group
Number analyzed (Participants) | 46 | 44 | 60
score on a scale
  Baseline | 7.6087 [7.0972 to 8.1201] | 7.6363 [7.0953 to 8.1774] | 6.5333 [6.1052 to 6.9615]
  1-year: number analyzed (Participants) | 39 | 40 | 45
  1-year | 6.1282 [5.3622 to 6.8942] | 6.6000 [5.8481 to 7.3519] | 6.3111 [5.8096 to 6.8126]
  3-years: number analyzed (Participants) | 36 | 35 | 39
  3-years | 5.5556 [4.7537 to 6.3574] | 6.0286 [5.3636 to 6.6935] | 5.6154 [5.1134 to 6.1174]
  7-years: number analyzed (Participants) | 36 | 36 | 34
  7-years | 4.8056 [4.2016 to 5.4095] | 5.6111 [4.9612 to 6.2611] | 5.4412 [4.9644 to 5.9179]
  10-12-years: number analyzed (Participants) | 35 | 28 | 30
  10-12-years | 4.6452 [4.0354 to 5.2549] | 5.2143 [4.5205 to 5.9080] | 5.1143 [4.5142 to 5.7143]
  15-years: number analyzed (Participants) | 26 | 21 | 30
  15-years | 4.1538 [3.4251 to 4.8826] | 4.8571 [4.1930 to 5.5213] | 5.0333 [4.5788 to 5.4878]
Statistical Analysis 1: Comparison: Low-tension vs High-tension vs Uninjured Control Group; These results are from the 15-year analysis; Test type: Superiority; p = .08, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were self-reported by subjects at each follow-up time-point beginning at 6 months and ending with the 15-year follow-up.
Description: Subjects reported injuries using a 'subsequent injuries survey.' There were no study related adverse events, as all events reported are expected surgical events.
Arm/Group | Low-tension | High-tension | Uninjured Control Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44 | 0/60
Other Adverse Events (participants affected / at risk) | 11/46 | 20/44 | 6/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-tension (N=46) | High-tension (N=44) | Uninjured Control Group (N=60)
contralateral ACL tear (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 1 (1)
Meniscal Tear (index) (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (10) | 2 (2)
Meniscal tear (contralateral) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
MCL Tear (index) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
MCL Tear (contralateral) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Other Knee Injury (index) (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1)
Other knee injury (contralateral) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (2)
Other knee injury (limb unspecified) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Graft Failure (Musculoskeletal and connective tissue disorders) | 2 (4) | 4 (4) | 0 (0)

LIMITATIONS AND CAVEATS:
The study participant retention rate dropped over time.

It should be noted that the method used to determine the Radiographic Joint Space Narrowing outcome measure changed overtime. To account for this, the baseline measure was determined with each method at each timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT00434837/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT00434837/ICF_002.pdf